CLINICAL TRIAL: NCT02728856
Title: Evaluation of the Irritation Potential of Products in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18598
Record Dates: First submitted 2016-03-03; First posted 2016-04-05 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sun Protection Factor (SPF) 50 Z15-034(BAY987516) (Experimental): Study staff will administer the control in one eye and a test sunscreen in the other eye according to the assigned randomization schedule.
  Interventions: Other: Sunscreen Spray SPF50 Z15-034(BAY987516); Other: Shampoo Control
- Sunscreen Spray SPF50 Z15-038(BAY987516) (Experimental): Study staff will administer the control in one eye and a test sunscreen in the other eye according to the assigned randomization schedule.
  Interventions: Other: Shampoo Control; Other: Sunscreen Spray SPF50 Z15-038(BAY987516)

INTERVENTIONS:
Other: Sunscreen Spray SPF50 Z15-034(BAY987516) — Study staff will administer the control in one eye and a test sunscreen in the other eye according to the assigned randomization schedule.
  Arms: Sun Protection Factor (SPF) 50 Z15-034(BAY987516)
Other: Shampoo Control — Study staff will administer the control in one eye and a test sunscreen in the other eye according to the assigned randomization schedule.
Other: Sunscreen Spray SPF50 Z15-038(BAY987516) — Study staff will administer the control in one eye and a test sunscreen in the other eye according to the assigned randomization schedule.
  Arms: Sunscreen Spray SPF50 Z15-038(BAY987516)

SUMMARY:
To evaluate the human eye irritation potential of two test sunscreen formulation

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy males or females between the ages of 18 to 60 years inclusive with no medical conditions of the eyes.
* Do not wear contact lenses or, if he/she does wear contact lenses, is willing to refrain from wearing these during the test period.
* Willing to report any medications taken during the study.
* Willing to have the test materials instilled into the eyes and follow all protocol requirements.
* Have been informed and have given written consent to participate in the study.

Exclusion Criteria:

* Has ocular disease or peri-orbital dermatitis or trauma, infections or chronic eye conditions that may affect the study outcome.
* Has systemic illness which affects the eyes, including diabetes, thyroid disease, sarcoidosis, hypertension, atherosclerosis, lupus, multiple sclerosis, sickle cell disease, acquired immune deficiency syndrome (AIDs), severer rheumatoid arthritis. results as determined by the investigator.
* Must not have a history of pre-existing sensitivity or other types of allergy to any eye products.
* Must not have received and used an Investigational New Drug within the thirty days immediately preceding the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2016-02-27 (Actual); Study Completion 2016-02-27 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of discomfort in the eyes assessed by 5 point scale | Up to 1 day
Intensity of Lacrimation assessed by 5 grading scale | Up to 1 day
Intensity of Bulbar Conjunctiva Irritation assessed by 4 grading scale | Up to 1 day
Intensity of Palpebral Conjunctiva Irritation assessed by 4 grading scale | Up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States